CLINICAL TRIAL: NCT05403996
Title: Effects of an Active Break Program at School on Physical Activity and On-task Behavior in Children From 6 to 12 Years Old
Brief Title: Effects of an Active Break Program at Primary School
Acronym: Activa-Mente
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de La Frontera (Other)
Collaborators: Playa Ancha University (Other); Universidad Metropolitana de Ciencias de la Educacion (Other)
Responsible Party: Principal Investigator, Nicolas Aguilar Farias, Phd, Universidad de La Frontera
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UPLA-005-2022
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Health Behavior; Behavior, Child
Keywords: physical activity; physical activity enjoyment; on-task behavior
MeSH Terms: conditions — Health Behavior; Child Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Pilot cluster randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activa-Mente (Intervention) (Experimental): The active break program involves the presentation of video (4.5 min) with moderate-to-vigorous physical activities. These active breaks will be performed 6 times per day during 6 weeks.
  Interventions: Behavioral: Activa-Mente
- Control group (No Intervention): This group of students will not be exposed to the intervention.

INTERVENTIONS:
Behavioral: Activa-Mente — Active break program
  Arms: Activa-Mente (Intervention)

SUMMARY:
The purpose of this study is to assess the effectiveness of an active break program at school on physical activity levels and enjoyment, and on-task behavior in children.

DETAILED DESCRIPTION:
The protocol will include third and fourth-grade students (children aged 8 to 10 years) from elementary schools in the Valparaíso Region, Chile. Four school classes from two schools (intervention and control school) will be included. The intervention school will carry out the active break program, ACTIVA-MENTE This program consists of the application of a 4-and-a-half-minute video with moderate to vigorous-intensity physical activity. These breaks will take place 6 times a day in classes for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren aged 8 to 10 years old (third to fourth grade of primary education).

Exclusion Criteria:

* Children with school attendance lower than 90 per cent (excluded from data analysis).
* Any medical condition that impedes physical activity breaks.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Physical activity | 6 weeks
  Physical activity will be measured with waist-worn ActiGraph GT3X+ accelerometers for seven days. Physical activity intensities will be derived from the accelerometer counts. Evenson cut points will be used to classify counts into physical activity intensities. Physical activity will be classified as light, moderate-to-vigorous and total physical activity.
On-task behavior | 6 weeks
  The Direct Behaviour Rating Scale will be used to measure on-task behavior at the individual level. This scale measures academically engaged, respectful and disruptive behavior. For each domain, the scale uses a per cent grading system in which 0% indicates 'never' while 100% indicates 'always'. At the group level, the Classroom Behaviour and Assets Survey will be used teachers who will be asked to indicate the proportion of the class displaying on-task behavior as defined by the individual behavior tool. Response options include: 0 (0 students), 1 (1-2 students), 2 (a few students), 3 (about ¼ of the class), 4 (about ½ of the class), 5 (about ¾ of the class), 6 (most of the class), and 7 (all of the class).

SECONDARY OUTCOMES:
Physical activity enjoyment | 6 weeks
  The Physical Activity Enjoyment Scale (PACES) will be used to measure enjoyment during the active breaks. Each of the 14 items of this instrument includes a Likert-type scale that ranges from 1 (Disagree a lot) to 5 (Agree a lot).

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Reyes, PhD, Principal Investigator — Playa Ancha University
Locations (1):
- Facultad de Ciencias de la Actividad Física y del Deporte, Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: Undecided
The anonymized and raw data supporting the conclusions of this study will be made available by the principal investigator, upon reasonable request.

REFERENCES:
- [Derived] Reyes-Amigo T, Grao-Cruces A, Sanchez-Oliva D, Garcia-Hermoso A, Reyes-Molina D, Yanez-Sepulveda R, Olivares-Arancibia J, Hurtado-Almonacid J, Paez-Herrera J, Salinas-Gallardo G, Mendoza E, Ovalle-Fernandez C, Sepulveda-Figueroa F, Ibarra-Mora J. Acute effect of school-based active breaks on physical activity level and on-task classroom behavior in primary schoolchildren. Front Public Health. 2025 Oct 30;13:1644819. doi: 10.3389/fpubh.2025.1644819. eCollection 2025. PMID 41246058
- [Derived] Reyes-Amigo T, Ibarra-Mora J, Aguilar-Farias N, Gomez-Alvarez N, Carrasco-Beltran H, Zapata-Lamana R, Hurtado-Almonacid J, Paez-Herrera J, Yanez-Sepulveda R, Cortes G, Rolle-Caceres G, Bezerra A. An active break program (ACTIVA-MENTE) at elementary schools in Chile: study protocol for a pilot cluster randomized controlled trial. Front Public Health. 2024 Jan 8;11:1243592. doi: 10.3389/fpubh.2023.1243592. eCollection 2023. PMID 38259740